CLINICAL TRIAL: NCT05354050
Title: A Phase 1 Single-center Pharmacokinetic Study of DARE-BV1 in Healthy Female Subjects
Brief Title: Pharmacokinetic Study of DARE-BV1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DARE-BV1-PK1
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DARE-BV1 (Experimental)
  Interventions: Drug: DARE-BV1

INTERVENTIONS:
Drug: DARE-BV1 — 2% Clindamycin 100 MG

SUMMARY:
Single-Center, Phase 1, Single-dose PK study of DARE-BV1 (2% clindamycin phosphate vaginal gel, 100mg) under development for the treatment of bacterial vaginosis (BV).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be females >= 18 years of age with no known medical conditions that, in the Investigator's opinion, may interfere with study participation.
2. Subjects may engage in heterosexual intercourse between Screening and Day-1, but must agree to abstain from sexual intercourse and/or sexual activity throughout the 7 days following treatment.
3. Subjects of childbearing potential should use adequate birth control between Screening and Day 1 if engaging in heterosexual intercourse, and should not plan on becoming pregnant for the duration of the study. Acceptable forms of birth control include oral contraceptives ("the pill"), intrauterine devices (IUDs), contraceptive implants under the skin, patches or injections, and non-polyurethane condoms (e.g., latex, polyisoprene) without spermicide. Subjects in same sex relationships, or monogamous relationships with vasectomized males, may also participate. Abstinence may also be acceptable, per the Investigator's judgment. Oral or transdermal hormonal contraceptives must be in use for 1 full cycle (e.g., 4 to 8 weeks) prior to study drug application. Injectable or implanted contraceptives (e.g., Depo-Provera, Nexplanon, or hormonal IUD) must have been injected/inserted at least 7 days prior to study drug application.
4. Subjects who are not of childbearing potential will not need a urine pregnancy test prior to dosing or at subsequent visits. Subjects are considered to be of non-child bearing potential if one of the following is satisfied:

   1. Postmenopausal for at least 1 year prior to the Screening Visit (Visit 1) (defined as amenorrheic for more than 1 continuous year), or
   2. Surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) at least 6 months before first dose, or
   3. Non-surgical permanent sterilization procedure performed at least 3 months prior to study drug application.
5. Subjects must be willing to refrain from the use of all intra-vaginal products (e.g., douches, feminine deodorant sprays, female condoms, spermicides, vaginal moisturizers or lubricants, tampons, vaginal birth control rings [e.g., NuvaRing®], and diaphragms) through the study or Study Exit/Early Discontinuation.

Exclusion Criteria:

1. Subjects with active BV, vulvovaginitis, or other active infectious causes of cervicitis, vaginitis, or vulvitis, based on the results of the thorough clinical assessments and testing as described above or genital lesions or ulcers consistent with HPV, Herpes simplex, syphilis, chancroid, etc.). Subjects with a history of genital herpes or condylomata who have been asymptomatic for at least 6 months may be considered for eligibility.
2. Potential subjects who are pregnant or are breastfeeding or, if of child-bearing potential, unwilling to practice acceptable means of birth control or abstinence during the study as described above.
3. Subjects with a vaginal, vulvar, or genitourinary condition that, according to the Investigator's judgment, may confound the interpretation of clinical assessments. This includes urinary tract infections requiring antibiotics.
4. Subjects with a history of regional enteritis, ulcerative colitis, or a history of Clostridium difficile-associated diarrhea.
5. Subjects with known current drug or alcohol abuse that could impact study compliance.
6. Subjects currently receiving or who have received antifungal or antibacterial therapy (systemic or intravaginal) within 14 days of the Screening Visit (Visit 1).
7. Subjects who have used any other investigational product within 30 days of the Screening Visit (Visit 1).
8. Subjects with HPV 16 or 18 at screening (performed on subjects >25 years old).
9. Subjects with known sensitivity to clindamycin phosphate or other lincosamides or any of the inactive ingredients in the study drug.
10. Subjects with a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with study participation or study treatment administration or could interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the Pharmacokinetics (PK) | 7 days
  Evaluate the PK of a single dose of DARE-BV1 in healthy female subjects by assessment of plasma and vaginal clindamycin concentrations

SECONDARY OUTCOMES:
Safety and Tolerability by evaluation of Treatment Emergent Adverse Events | 21 days
  Assess the safety and tolerability of DARE-BV1 by looking at TEAEs & local site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mauck, MD, Study Director — Dare Bioscience, Inc.
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No